CLINICAL TRIAL: NCT05237947
Title: Single-Dose HPV Vaccination Among Young Adult Women in Costa Rica: the PRISMA-ESCUDDO Trial (PRevencIón Del Cáncer Cervical Con Una Sola Dosis de Vacuna Contra VPH en Mujeres Adultas Jóvenes)
Brief Title: Single-Dose HPV Vaccination for the Prevention of Cervical Cancer in Young Adult Women in Costa Rica, The PRISMA ESCUDDO Trial
Acronym: PRISMA
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: NCI-2022-00343; NCI-2022-00343 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); DCEG ERP 22G001-01; CEC-FUNIN-007-2021; 154376 (Other: National Cancer Institute)
Record Dates: First submitted 2022-02-08; First posted 2022-02-14 (Actual); Last update posted 2025-09-05 (Actual); Status verified 2025-09

CONDITIONS: Human Papillomavirus-Related Cervical Carcinoma
MeSH Terms: interventions — Diphtheria Toxoid; adacel; Diphtheria-Tetanus-acellular Pertussis Vaccines; Tetanus Toxoid; human papillomavirus vaccine, L1 type 16, 18; Human Papillomavirus Recombinant Vaccine nonavalent

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Arm I (Gardasil 9) (Experimental): Patients receive one dose of Gardasil 9 IM.
  Interventions: Other: Questionnaire Administration; Biological: Recombinant Human Papillomavirus Nonavalent Vaccine
- Arm II (Cervarix) (Experimental): Patients receive one dose of Cervarix IM.
  Interventions: Other: Questionnaire Administration; Biological: Recombinant Human Papillomavirus Bivalent Vaccine
- Arm III (Adacel) (Active Comparator): Patients receive one dose of Adacel IM.
  Interventions: Biological: Diphtheria Toxoid/Tetanus Toxoid/Acellular Pertussis Vaccine Adsorbed; Other: Questionnaire Administration

INTERVENTIONS:
Biological: Diphtheria Toxoid/Tetanus Toxoid/Acellular Pertussis Vaccine Adsorbed — Given IM
  Other Names: Adacel; Daptacel; Diphtheria and Tetanus Toxoids and Acellular Pertussis Vaccine Adsorbed; Diphtheria Toxoid Tetanus Toxoid Acellular Pertussis Vaccine Adsorbed; Diphtheria Toxoid/Tetanus Toxoid/Acellular Pertussis Vaccine; DTaP; Infanrix; Tripedia
  Arms: Arm III (Adacel)
Other: Questionnaire Administration — Ancillary studies
Biological: Recombinant Human Papillomavirus Bivalent Vaccine — Given IM
  Other Names: Cervarix; GSK-580299; HPV 16/18 L1 VLP/AS04 VAC; HPV-16/18 VLP/AS04 Vaccine; Human Papillomavirus 16/18 L1 Virus-Like Particle/AS04 Vaccine; Human Papillomavirus Bivalent Types 16 and 18 Vaccine, Recombinant; Human Papillomavirus Vaccine L1 16,18; Human Papillomavirus Vaccine, L1 Type 16, 18; Recombinant HPV Bivalent Vaccine
  Arms: Arm II (Cervarix)
Biological: Recombinant Human Papillomavirus Nonavalent Vaccine — Given IM
  Other Names: Gardasil 9; Nonavalent HPV VLP Vaccine; Recombinant HPV Nonavalent Vaccine; Recombinant Human Papillomavirus 9-valent Vaccine
  Arms: Arm I (Gardasil 9)

SUMMARY:
This phase IV trial tests whether a single dose of the human papillomavirus (HPV) vaccine works in preventing cervical cancer in young women in Costa Rica. Human papilloma viruses, called HPV, are a group of viruses that very frequently cause infection in both men and women, mainly in the genital organs. There are many types of HPV, and some can cause cancer. The World Health Organization recommends a two-dose schedule for adolescents 9-14 and three doses for individuals 15 years old or older. This study examines whether a single dose of HPV vaccine can reduce the frequency with which women between ages 18-30 become infected with HPV.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate one dose of nonavalent human papillomavirus (HPV) vaccination compared to no vaccination in the protection against incident HPV16/18 cervical HPV infections that persist 6-months or more in women aged 18 to 30 years who are cervical HPV16/18 deoxyribonucleic acid (DNA) negative prior to and at the time of vaccination.

II. To evaluate one dose of bivalent HPV vaccination compared to no vaccination in the protection against incident HPV16/18 cervical HPV infections that persist 6-months or more in women aged 18 to 30 years who are cervical HPV16/18 DNA negative prior to and at the time of vaccination.

SECONDARY OBJECTIVES:

I. To quantitate the benefit of one dose of HPV vaccination compared to no vaccination in the protection against incident HPV16/18 cervical HPV infections that persist 6-months or more in women aged 18 to 30 years regardless of cervical HPV DNA status at the time of vaccination.

II. To estimate the health impact of older-age single-dose HPV vaccination by modeling the number of cervical cancer cases prevented as well as the cost-effectiveness of cervical cancer prevention strategies incorporating vaccination and screening in Costa Rica.

III. To evaluate the immunogenicity (absolute levels and stability of serum antibodies) of single dose HPV vaccination in women.

IV. For each vaccine separately, to evaluate one dose of HPV vaccination compared to no vaccination in the protection against:

IVa. Any new HPV16/18 anal infection that persists 6+ months. IVb. Any new HPV16/18 oral infection that persists 6+ months. IVc. Any new carcinogenic HPV cervical, anal or oral infection detected at a single timepoint and that persists 6+ months.

IVd. Any new cervical HPV6/11 infection that persists 6+ months.

OUTLINE: Patients are randomized to 1 of 3 arms.

ARM I: Patients receive one dose of recombinant human papillomavirus nonavalent vaccine (Gardasil 9) intramuscularly (IM).

ARM II: Patients receive one dose of recombinant human papillomavirus bivalent vaccine (Cervarix) IM.

ARM III: Patients receive one dose of diphtheria toxoid/tetanus toxoid/acellular pertussis vaccine adsorbed vaccine (Adacel) IM.

After completion of study, patients are followed up at 6 and 12 months, and then every 6 months thereafter.

ELIGIBILITY:
Inclusion Criteria:

* INCLUSION CRITERIA AT ENROLLMENT: Female.
* INCLUSION CRITERIA AT ENROLLMENT: Aged between 18 and 30 years inclusive.
* INCLUSION CRITERIA AT ENROLLMENT: Living in the study area.
* INCLUSION CRITERIA AT ENROLLMENT: Able to communicate with study personnel.
* INCLUSION CRITERIA AT ENROLLMENT: Willing to participate in the study and sign the informed consent.
* INCLUSION CRITERIA AT ENROLLMENT: In good health as determined by a medical history (physical exam will be conducted if necessary per the doctor's criterion.
* DEFERRAL CRITERIA AT ENROLLMENT VISIT: The enrollment visit will be deferred (i.e., rescheduled for another date) for participants if: the self-collected cervical sample is not able to be collected.
* DEFERRAL CRITERIA AT THE VACCINATION VISIT: The vaccination visit will be deferred (i.e., rescheduled for another date) for participants if:

  * They have an acute disease that precludes vaccination (though vaccines can be administered to potential participants with a minor illness such as diarrhea and mild upper respiratory infection)
  * They are receiving immunosuppressive treatment, e.g. corticosteroids
  * They have received any registered vaccine in the last 15 days.

Exclusion Criteria:

* EXCLUSION CRITERIA AT ENROLLMENT VISIT: They have been vaccinated against human papillomavirus (HPV).
* EXCLUSION CRITERIA AT ENROLLMENT VISIT: They are allergic to yeast or another vaccine components.
* EXCLUSION CRITERIA AT ENROLLMENT VISIT: They have a diagnosis of an autoimmune, degenerative, or neurological disease without treatment or adequate control; a progressive or severe neurological disease; a genetic immunodeficiency; or any other serious chronic disease without treatment and / or adequate control that, according to the principal investigator or designee, for which vaccination is contraindicated.
* EXCLUSION CRITERIA AT ENROLLMENT VISIT: They have plans to move outside the country in the next six months.
* EXCLUSION CRITERIA AT ENROLLMENT VISIT: They refuse or are unable to self-collect the cervical sample.
* EXCLUSION CRITERIA AT ENROLLMENT VISIT: They are pregnant.
* EXCLUSION CRITERIA AT ENROLLMENT VISIT: They do not have an identification document.
* EXCLUSION CRITERIA AT ENROLLMENT VISIT: The clinician determining eligibility in agreement with the principal investigator considers that there is a reason that precludes participation.
* EXCLUSION CRITERIA AT VACCINATION VISIT: Between the enrollment and vaccine visit, they have been vaccinated against HPV.
* EXCLUSION CRITERIA AT VACCINATION VISIT: Between the enrollment and vaccine visit, they are being evaluated for or have received a diagnosis of: an autoimmune, degenerative, or neurological disease without treatment or adequate control; a progressive or severe neurological disease; a genetic immunodeficiency; or any other serious chronic disease without treatment and/or adequate control, for which vaccination is contraindicated according to the principal investigator or designee.
* EXCLUSION CRITERIA AT VACCINATION VISIT: They have plans to move outside the country in the next six months.
* EXCLUSION CRITERIA AT VACCINATION VISIT: They refuse the urine pregnancy test.
* EXCLUSION CRITERIA AT VACCINATION VISIT: They have a positive urine pregnancy test result.
* EXCLUSION CRITERIA AT VACCINATION VISIT: They are pregnant.
* EXCLUSION CRITERIA AT VACCINATION VISIT: They refuse or are unable to perform the self-collected cervical sample.
* EXCLUSION CRITERIA AT VACCINATION VISIT: The clinician determining eligibility in agreement with the principal investigator considers that there is a reason that precludes participation.

Ages: 18 Years to 30 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 5000 (Estimated)
Dates: Start 2022-03-01 (Actual); Primary Completion 2026-05-31 (Estimated); Study Completion 2026-05-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of persistent HPV infection | 6-month persistence observed during follow-up
  Will estimate the rate of incident persistent infections (i.e. the primary endpoint defined above) in each of the three arms of an ATP cohort and then estimate the two Vaccine Efficacies (VE), comparing each HPV vaccine arm against the control arm. Will require a one-sided p-value of < 0.0125 for statistical significance. The 97.5% confidence intervals for the VE will be calculated by inverting appropriate hypotheses tests.

SECONDARY OUTCOMES:
Benefit of one dose of HPV vaccination compared to no vaccination | 6-month persistence observed during follow-up
  Will require a one-sided p-value of < 0.0125 for statistical significance. The 97.5% confidence intervals for the VE will be calculated by inverting appropriate hypotheses tests.
Health impact of older-age single-dose HPV vaccination | 6-month persistence observed during follow-up
  Will require a one-sided p-value of < 0.0125 for statistical significance. The 97.5% confidence intervals for the VE will be calculated by inverting appropriate hypotheses tests.
Immunogenicity (absolute levels and stability of serum antibodies) of single dose HPV vaccination | 6-month persistence observed during follow-up
  Will report the Geometric Mean Titer (GMT) of the antibodies for each HPV type at the five follow-up visits.
New HPV16/18 anal infection | 6-month persistence observed during follow-up
  Will report the VE against any new carcinogenic HPV type and against HPV 6/11 in the according to protocol (ATP) cohort using an analysis plan similar to that described for the primary objectives.
New HPV16/18 oral infection | 6-month persistence observed during follow-up
  Will report the VE against any new carcinogenic HPV type and against HPV 6/11 in the according to protocol (ATP) cohort using an analysis plan similar to that described for the primary objectives.
Carcinogenic HPV cervical, anal or oral infection detected at a single timepoint | 6-month persistence observed during follow-up
  Will report the VE against any new carcinogenic HPV type and against HPV 6/11 in the according to protocol (ATP) cohort using an analysis plan similar to that described for the primary objectives.
Cervical HPV6/11 infection | 6-month persistence observed during follow-up
  Will report the VE against any new carcinogenic HPV type and against HPV 6/11 in the according to protocol (ATP) cohort using an analysis plan similar to that described for the primary objectives.

CONTACTS AND LOCATIONS:
Overall Officials: Aimee R Kreimer, Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- Agencia Costarricense de Investigaciones Biomédicas (ACIB), Liberia, Guanacaste Province, Costa Rica

REFERENCES:
- [Derived] Bergman H, Henschke N, Arevalo-Rodriguez I, Buckley BS, Crosbie EJ, Davies JC, Dwan K, Golder SP, Loke YK, Probyn K, Petkovic J, Villanueva G, Morrison J. Human papillomavirus (HPV) vaccination for the prevention of cervical cancer and other HPV-related diseases: a network meta-analysis. Cochrane Database Syst Rev. 2025 Nov 24;11(11):CD015364. doi: 10.1002/14651858.CD015364.pub2. PMID 41276263